CLINICAL TRIAL: NCT06196320
Title: Tenecteplase Reperfusion Therapy in Acute Ischaemic Cerebrovascular Events-5 Improving Neurological Functional Outcomes in Basilar Artery Occlusion With Tenecteplase in Extended Time Window: Multicentre, Prospective, Open-label, Blinded Endpoint (PROBE), Phase 3, Randomized Controlled Trial
Brief Title: Tenecteplase Reperfusion Therapy in Acute Ischaemic Cerebrovascular Events-5
Acronym: TRACE-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSA2023YJ002
Record Dates: First submitted 2023-12-06; First posted 2024-01-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke, Acute
Keywords: rhTNK-tPA; rt-PA; Ischemic stroke; phase III trial; basilar artery occlusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; TNK-tissue plasminogen activator; Practice Guidelines as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenecteplase (Experimental): Intravenous tenecteplase (0.25mg/kg, maximum 25mg) within 24 hours ± thrombectomy at treating clinician's discretion
  Interventions: Drug: Tenecteplase
- Best Practice (which may include intravenous Alteplase) (Active Comparator): Intravenous alteplase (0.9mg/kg) within 4.5 hours from stroke onset or standard care (no lysis) ± thrombectomy at treating clinician's discretion
  Interventions: Drug: Best Practice (which may include intravenous Alteplase)

INTERVENTIONS:
Drug: Tenecteplase — Intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over 5-10 seconds) within 24 hours ± thrombectomy at treating clinician's discretion
  Other Names: rhTNK-tPA; TNK-tPA
  Arms: Tenecteplase
Drug: Best Practice (which may include intravenous Alteplase) — Intravenous alteplase (0.9mg/kg) within 4.5 hours from stroke onset or standard care (no lysis) ± thrombectomy at treating clinician's discretion
  Other Names: rt-PA
  Arms: Best Practice (which may include intravenous Alteplase)

SUMMARY:
The trial is a multicentre, prospective, open-label, blinded endpoint (PROBE), phase 3, randomized controlled design. Patients with acute ischemic stroke due to basilar artery occlusion presenting within 24 hours will be randomized 1:1 to intravenous tenecteplase (0.25mg/kg, maximum 25mg) ± thrombectomy or 'best practice'which may be alteplase (0.9mg/kg) within 4.5 hours from stroke onset or standard care (no lysis) ± thrombectomy at treating clinician's discretion.

DETAILED DESCRIPTION:
The study will be a multicentre, prospective, open-label, blinded endpoint (PROBE), randomized controlled trial (2 arm with 1:1 randomization) in patients with acute ischemic stroke due to basilar artery occlusion presenting to hospital within 24 hours of symptom onset.

Patients will be required to have complete or near-complete occlusion of the basilar artery on baseline computed tomography angiography (CTA)/magnetic resonance angiography (MRA), defined as 'potentially retrievable' thrombus in the basilar artery. Thrombectomy is permitted within 24 hours as part of standard care but is not mandatory.

Patients will be randomized to treatment with either standard of care (no intravenous thrombolytic treatment or intravenous alteplase 0.9mg/kg within 4.5 hours from stroke onset) or intravenous tenecteplase (0.25mg/kg, maximum 25mg). Time of onset of symptoms is defined as described by the patient or witness; if unknown, it is considered to be the last time the patient was seen well. In patients presenting with mild (e.g. vertigo, dizziness, headache, diplopia, dysarthria) stuttering symptoms followed by sudden onset of clinical deterioration with decrease in conscious state or moderate to severe motor deficits, the time of deterioration in clinical state is taken as the estimated time of basilar artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.
2. Patients presenting with posterior circulation ischemic stroke symptoms due to near-complete or complete basilar artery occlusion within 24 hours from symptom onset (or clinical deterioration/coma) or the time the patient was last known to be well.
3. Presence of a basilar artery occlusion, proven by CT Angiography or MR Angiography. Basilar artery occlusion will be defined as 'potentially retrievable' occlusion at the basilar artery. This can be a near or complete occlusion.
4. Premorbid mRS ≤3 (independent function or requiring only minor domestic assistance and able to manage alone for at least 1 week).
5. Local legal requirements for consent have been satisfied.

Exclusion Criteria:

1. Intracerebral haemorrhage (ICH) or other diagnosis (e.g. tumour) identified by baseline imaging.
2. Posterior circulation Acute Stroke Prognosis Early CT Score (PC-ASPECTS) <6 on non-contrast CT (NCCT) or CTA-source images or MRI diffusion weighted imaging (DWI).
3. Significant cerebellar mass effect or acute hydrocephalus.
4. Established frank hypodensity on non-contrast CT indicating subacute infarction.
5. Bilateral extensive brainstem ischemia.
6. Pre-stroke mRS of ≥4 (indicating moderate to severe previous disability).
7. Other standard contraindications to intravenous thrombolysis.
8. Contraindication to imaging with contrast agents.
9. Clinically evident pregnant women.
10. Vessel imaging showing both anterior and posterior circulation large vessel occlusion.
11. Current participation in another research drug treatment protocol.
12. Known terminal illness such that the patients would not be expected to survive a year.
13. Planned withdrawal of care or comfort care measures.
14. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) 0-1 or return to baseline mRS | 3 months
  The proportion of patients with Modified Rankin Scale (mRS) 0-1 (no disability) or return to baseline mRS (if baseline premorbid mRS =2-3) at 3 months. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) 0-2 or return to baseline mRS | 3 months
  Proportion of patients with Modified Rankin Scale (mRS) 0-2 or return to baseline mRS at 3 months. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Modified Rankin Scale (mRS) 0-3 or return to baseline mRS | 3 months
  Proportion of patients with Modified Rankin Scale (mRS) 0-3 or return to baseline mRS at 3 months. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Ordinal analysis of the Modified Rankin Scale (mRS) | 3 months
  Ordinal analysis of the Modified Rankin Scale (mRS), merging category 5-6, at 3 months. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Early neurological improvement | 72 hours
  Proportion of patients achieving early clinical improvement (reduction in acute - 72 hour National Institutes of Health Stroke Scale [NIHSS] score of ≥8 or 72 hour NIHSS 0-1).
Successful reperfusion | initial DSA run prior to thrombectomy
  Proportion of patients with complete occlusion at baseline who achieve expanded Thrombolysis In Cerebral Infarction score (eTICI) 2b/3 on initial digital subtraction angiography (DSA) run prior to thrombectomy.
Symptomatic intracranial hemorrhage (sICH) | 36 hours
  Proportion of patients with symptomatic intracranial hemorrhage (sICH) defined as local or remote parenchymal hemorrhage type 2 (PH2) on the 22-36 hours post-treatment imaging scan, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline, or from the lowest NIHSS value between baseline and 24 hours, or leading to death.
All-cause mortality | 90 days
  All-cause mortality within 90 days.
Severe disability or death | 90 days
  Proportion of patients with Modified Rankin Scale (mRS) 5-6 at 90 days (severe disability or death). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Clinical deterioration | 24 hours
  Proportion of patients with partially occlusive thrombus at baseline who have clinical deterioration within 24 hours leading to further treatment (e.g. endovascular thrombectomy).
Vessel recanalization | 24+/-6 hours
  Vessel recanalization rate evaluated by CT or MR angiography within 24+/-6 hours (if performed).

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital; Bruce Campbell, MD, PhD, Principal Investigator — University of Melbourne; Fana Alemseged, MD, PhD, Study Director — University of Melbourne; Yunyun Xiong, MD, PhD, Study Director — Beijing Tiantan Hospital
Locations (59):
- China (59):
  - Taihe County Traditional Chinese Medicine Hospital, Fuyang, Anhui
  - Lixin County People's Hospital, Haozhou, Anhui
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - First People's Hospital of Tianshui, Tianshui, Gansu
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Heyuan People's Hospital, Heyuan, Guangdong
  - Huazhou People's Hospital, Huazhou, Guangdong
  - Shaoguan Qujiang District People's Hospital, Shaoguan, Guangdong
  - The Second Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second People's Hospital of Guiyang, Guiyang, Guizhou
  - Qiandongnanzhou People's Hospital, Qiandongnan, Guizhou
  - Haikou People's Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Qiu County People's Hospital, Handan, Hebei
  - The Second Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Tangshan Guye Traditional Chinese Medicine Hospital, Tangshan, Hebei
  - Qinghe County People's Hospital, Xingtai, Hebei
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Hongxinglong Hospital of Beidahuang Group, Shuangyashan, Heilongjiang
  - Huaxian People's Hospital of Henan, Anyang, Henan
  - Jiaozuo Coal Industry Central Hospital, Jiaozuo, Henan
  - The First People Hospital of Lingbao, Lingbao, Henan
  - Liuyang Jili Hospital, Liuyang, Henan
  - Nanshi Hospital of Nanyang, Nanyang, Henan
  - Nanle County People's Hospital, Puyang, Henan
  - Nanle Zhongxing Hospital, Puyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Guangshan County People's Hospital, Xinyang, Henan
  - Xi County People's Hospital, Xinyang, Henan
  - Taikang Xian People's Hospital, Zhoukou, Henan
  - People's Hospital of Queshan, Zhumadian, Henan
  - Zhumadian Traditional Chinese Medicine Hospital, Zhumadian, Henan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - The Fourth People's Hospital of Chenzhou, Chenzhou, Hunan
  - Hengyang Central Hospital, Hengyang, Hunan
  - Keshketeng Banner Chinese-Mongolian Hospital, Keshketeng Banner, Inner Mongolia
  - Tongliao People's Hospital, Tongliao, Inner Mongolia
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - Jilin Electric Power Hospital, Changchun, Jilin
  - Siping City Central People's Hospital, Siping, Jilin
  - Liuhe County People's Hospital, Tonghua, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The Second People's Hospital of Dongying, Dongying, Shandong
  - Gaomi People's Hospital, Gaomi, Shandong
  - Laizhou City People's Hospital, Laizhou, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - The Second Affiliated Hospital of Shandong First Medical University, Taian, Shandong
  - The Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Yantai Taochun Central Hospital, Yantai, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Linfen Central Hospital, Linfen, Shanxi
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Beilun District People's Hospital, Ningbo, Zhejiang
  - Beijing Daxing District People's Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiong Y, Alemseged F, Cao Z, Schwamm LH, Zhang S, Parsons MW, Fisher M, Hao Y, Jin A, Yin J, Jiang Y, Che F, Wang L, Zhou L, Dai H, Zhao Y, Duan C, Wu S, Feng G, Zong L, Ye W, Wang Z, Xu Z, Wang H, Hao M, Ma Y, Meng X, Li H, Li Z, Wang Y, Liu L, Zhao X, Campbell BCV, Wang Y; TRACE-5 investigators. Tenecteplase versus standard medical treatment for basilar artery occlusion within 24 h (TRACE-5): a multicentre, prospective, randomised, open-label, blinded-endpoint, superiority, phase 3 trial. Lancet. 2026 Feb 5:S0140-6736(25)02633-9. doi: 10.1016/S0140-6736(25)02633-9. Online ahead of print. PMID 41655588
- [Derived] Xiong Y, Alemseged F, Cao Z, Schwamm LH, Parsons M, Fisher M, Wu S, Campbell BCV, Wang Y. Tenecteplase versus standard care in patients with acute basilar artery occlusion: a multi-centre, prospective, randomised, open-label, blinded endpoint, phase 3, controlled trial. Stroke Vasc Neurol. 2025 Oct 28:svn-2025-004432. doi: 10.1136/svn-2025-004432. Online ahead of print. PMID 41151803